CLINICAL TRIAL: NCT01238471
Title: Oral Propranolol Versus Placebo for Early Stages of Retinopathy of Prematurity (ROP): A Pilot, Randomized and Prospective Study.
Brief Title: Oral Propranolol Versus Placebo for Early Stages of Retinopathy of Prematurity: A Randomized and Prospective Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Hadassah Medical Organization (Other); Laniado Hospital (Other); Nazareth Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0479-09CTIL; Israeli Health Ministry (Other: 1764/2117 Israeli Health Ministry Pharmaceutical Administration)
Record Dates: First submitted 2010-11-08; First posted 2010-11-10 (Estimated); Results first posted 2014-06-10 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Retinopathy of Prematurity
Keywords: retinopathy of prematurity; Propranolol; Vascular endothelial growth factor; premature infant
MeSH Terms: conditions — Retinopathy of Prematurity; Premature Birth | interventions — Propranolol; Adrenergic beta-Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propranolol (Experimental): Oral propranolol for premature infants allocated to this arm by randomization
  Interventions: Drug: propranolol
- Oral sucrose 5% (Placebo Comparator): Placebo: Oral sucrose 5% for premature infants allocated to control arm by randomization
  Interventions: Drug: sucrose 5%

INTERVENTIONS:
Drug: propranolol — 2 mg per kg per day divided in 3 doses for 2-4 weeks
  Other Names: beta blocker; deralin
  Arms: Propranolol
Drug: sucrose 5% — 2 ml per Kg per day divided in 3 doses for 2-4 weeks
  Other Names: sucrose sugar
  Arms: Oral sucrose 5%

SUMMARY:
In premature infants, propranolol (Prop) treatment might suppress continuing neo-vascularization (NV) and decelerate the progression of retinopathy of prematurity (ROP) towards its severe stages (III-V), thus avoiding the need of interventions (CRYO and/or LASER photo-coagulation of the ischemic retina and preventing severe ocular sequelae. We therefore plan to prospectively investigate the influence of prop versus placebo in VLBW infants with ROP stage 1 (zone I), with stage 2 or higher (any zone) or with Plus disease, along with close follow up regarding safety of prop administration and its effect on ROP.

DETAILED DESCRIPTION:
Retinopathy of prematurity (ROP) affects the retinal microvasculature, mostly of very-low-birth-weight (VLBW: < 1500g) premature infants, and is a significant complication of extreme prematurity leading sometimes to devastating consequences. Although ROP is usually mild with no harm, it happens not very rarely to be aggressive causing neo-vascularization (NV) in the immature retina that at times can progress to severe fibrovascular proliferation, retinal detachment and blindness (1). Major risk factors for ROP are low gestational age, low birth weight, hyperoxia, respiratory distress syndrome (RDS) and intraventricular hemorrhage (IVH) (2) as well as postnatal steroid therapy (3). Of note is one report showing that the use of beta-blocking agents by the mother before birth was found to be associated with the development of ROP (4). However, so far no one reported a similar effect of the postnatal use of beta blockers on ROP.

The incidence of ROP is inversely related to gestational age (GA) and birth weight (BW). The condition develops in 51% of infants with a birth weight (BW) <1700 g (5). In infants weighing less than 1250 g, 50% show some evidence of ROP and 10% progress to stage III ROP. According to the Israeli VLBW-Database in 2007, 23.9% of infants develop ROP (all stages), while 4.8% develop severe ROP (stage III-IV) (4). Worldwide, at least 50,000 children are blind from ROP (2,7). In South Africa it accounts for 10.6% of cases of childhood blindness (8). In the US, annually, 500-700 children become blind due to ROP, and 2100 infants will be affected by cicatricial sequelae, such as myopia, strabismus, as well as late-onset retinal detachment (1).

LASER photocoagulation of the ischemic retina is the therapy of choice for moderate to severe ROP and is required in 19.8%, 7.7%. 1.5% and 0.6% of infants weighing 500-749g, 750-999g, 1000-1249g, 1250-1499g, respectively (2). In Israel, 4% of VLBW infants needed LASER photocoagulation or cryo therapy during 2007 (6).

The pathogenesis of ROP is multifactorial and two pathogenetic theories have been proposed:

(A) One-phase theory: Mesenchymal spindle cells when exposed to extrauterine hyperoxia, develop gap junctions that interfere with normal vascular formation and trigger a neovascular response (9).

(B) Two-phase theory: The first phase (hyperoxic phase, vaso-obliterative), consists of retinal vasoconstriction and irreversible capillary endothelial cell damage. As the retinal area that is supplied by the affected vessels becomes ischemic, angiogenic factors, such as vascular endothelial growth factor (VEGF) are produced by mesenchymal spindle cells in that ischemic retina to provide neo vascularization (NV) channels (second phase, vaso-proliferative)(10).

Increasing evidence supports the key role of VEGF in the pathogenesis of ROP, wherein VEGF is down-regulated in the vaso-obliterative first phase and up-regulated in the vaso-proliferative second phase (11). Numerous studies have been performed in an animal model of oxygen-induced retinopathy (OIR), wherein newborn rats, mice, kitten and beagle puppies were exposed to 75-100% O2 for 5 days starting at day 7 of life (11). ROP usually develops in 100% of the O2-exposed rats (12).

The expression of various angiogenetic and inflammation genes has been studied in oxygen-induced retinopathy (OIR). Sato et al (13) investigated the expression of 94 genes in OIR using microarray analysis and reverse transcriptase-polymerase chain reaction (RT-PCR). They observed that: (a) Inflammation genes were up-regulated at days 12-13 of life when the degree of both central avascular area and central vasoconstriction were maximal; this up-regulation continued until day 21 of life; (b) Extra retinal vascularization was most noticeable at days 16-17 of life, when angiogenesis genes (VEGF-A, angiopoietin-2) were at their highest expression.

There is also increasing evidence of up-regulation of VEGF by sympathomimetic agents. In this regard, norepinephrine has been shown to stimulate myocardial angiogenesis in rats (14). In cultured retinal endothelial cells, Steinle et al (15) showed that significantly increased expression of beta-3 receptors could promote migration and proliferation (two markers of angiogenic phenotype) of retinal endothelial cells.

In addition, in cancer cell cultures, catecholamines (norepinephrine and epinephrine) induced an increase of VEGF expression in a tissue culture of nasopharyngeal carcinoma, an effect that was blocked by propranolol (prop) (a non-selective beta blocker) (16). Evidence exists for norepinephrine-induced invasiveness with increased VEGF in human pancreatic cell lines, could also be blocked by prop (17). Blockade of these effects by prop raised the prospects of a possible chemo-prevention of vascularization-rich tumors by propranolol.

Recent studies have shown that administration of beta-blockers (both locally and systemic) can mitigate NV, probably by down regulation of VEGF. In an animal model of OIR, topical timolol (a beta blocker) prevented the development of OIR in 40% of rats and mitigated the severity of OIR in the remaining 60% of rats that had developed OIR (12,18). In addition, timolol had a protective effect, whereby NV occurred in 65% of timolol-treated as compared to 100% NV in untreated rats (19). Furthermore, VEGF expression was lower in timolol-treated rats than in controls (room air). In contrast, Zheng et al (20) found no effect of prop on the VEGF protein and on messenger ribonucleic acid (mRNA) expression in the retina of diabetic rats with retinopathy.

ROP and infantile hemangiomas (a rather common phenomena in premature infants) supposedly share the same pathogenetic role of angiogenic factors such as VEGF (21). In a recent report by Praveen et al (22), a possible association between ROP and infantile hemangiomas at discharge was studied in premature infants weighing <1250 g. Infantile hemangiomas were found to be independently associated with any stage of ROP: infantile hemangiomas were present in 16.8% of neonates with ROP as compared with 6.7% of those without ROP. However, neither the size nor the number of infantile hemangiomas showed any association with the severity of ROP.

The above-mentioned published findings point to a VEGF-mediated pathogenesis of both ROP and infantile hemangiomas, wherein VEGF expression is reportedly up-regulated by sympathomimetic agents and blocked by beta blockers. Furthermore, on the clinical scene, the usefulness of prop in mitigating the progression of infantile hemangiomas has been recently reported (23-32). Infants with severe or life-threatening hemangiomas were successfully treated with prop, with no adverse effects. One potential explanation for the effect of prop on hemangiomas includes: (a) vasoconstriction, or (b) decreased expression of VEGF and basic fibroblast growth factor (bFGF) genes through the down-regulation of RAF-mitogen-activated protein kinase pathway (33) (which explains the progressive improvement of hemangioma), or (c) a triggering of capillary endothelial cells apoptosis (34).

Prop administration has been observed to be safe in infants and toddlers (23-32, 35). Love et al (35) found that after 40 years of clinical use in infants and toddlers, there is no documented case of death or serious cardiovascular disease as a direct result of exposure to beta-blockers. Furthermore, prop was also reported to be safe when given to premature infants for treatment of neonatal thyrotoxicosis, neonatal arrhythmia or life-threatening hemangioma (32, 36-39). In five extreme-low-birth weight infants (weight <1000 g), the use of prop for neonatal thyrotoxicosis was beneficial and had no adverse effects (36). The safety of prop use was also reported in a 34-week infant (37) and a for 37-week infant (38) with thyrotoxicosis, and also in a 35-week infant with neonatal arrhythmia (39). Furthermore, a 28-week premature infant was treated for18 weeks with prop for a thoracic hemangioma without untoward effects (32).

ELIGIBILITY:
Inclusion Criteria:

Evidence for ROP that might progress and that includes any one of the following:

* Stage 1 (zone I)
* Stage 2 or higher (zones I, II or III), or Plus disease. The classification of ROP is according to International Classification of Retinopathy of Prematurity (ICROP) 2005 (40) (Appendix I, with scheme of retina showing zones and clock hours).Zone III ROP is not included since it will always regress spontaneously.

Exclusion Criteria:

* The presence of one or more of the following conditions at enrollment in the study:
* More than 10 episodes of bradycardia of prematurity/day (HR< 90 bpm) [
* Atrio-ventricular (A-V) block [2nd or 3rd degree]
* Significant congenital heart anomaly [not including patent ductus arteriosus, patent foramen ovale or small ventricular septal defect]
* Heart failure
* Hypotension (mean blood pressure <45 mmHg)
* Hypoglycemia (<50mg/dL)
* Platelet count <100000/mm3

Ages: 4 Weeks to 14 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2010-05; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Israel (4):
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Organization, Jerusalem
  - Nazareth Hospital, Nazareth
  - Laniado Hospital, Netanya

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Propranolol | Oral Sucrose 5%
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propranolol | Oral Sucrose 5% | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: days] | 60.9 (4.9) | 64.4 (10.5) | 62.6 (7.7)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 10 | 20
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  Israel | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Regression of Retinopathy of Prematurity (ROP) in Premature Infants by Propranolol Therapy
Description: If ROP regresses without the need for treatment (laser and/or CRYO), this will be considered a favorable outcome. On the other hand, if ROP progresses to require treatment, it will be regarded as an unfavorable outcome.
  Evidence for regression of ROP was observed by serial retinal examinations performed by ophthalmologists as well as by reduction for the need of invasive interventions such as laser photocoagulation of disease areas in the retina.
Time Frame: propranolol therapy for up 4 weeks
Measure: Number; unit: cases
Arm/Group | Propranolol | Oral Sucrose 5%
Number analyzed (Participants) | 10 | 10
cases | 4 | 8

2. Secondary Outcome: Safety of Propranolol Therapy in Premature Infants
Description: Close monitoring for possible side effects of propranolol in premature infants
Time Frame: 4 weeks of propranolol therapy in premature infants
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Propranolol | Oral Sucrose 5%
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propranolol (N=10) | Oral Sucrose 5% (N=10)
bradycardia (Cardiac disorders) | 0 (0) | 0 (0) — none had bradycardia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other